CLINICAL TRIAL: NCT05036460
Title: Real-time Sonography as an Auxiliary Approach to Detect Inadvertent Esophageal Intubation Before Ventilation Among Suspected Difficult Intubation Patients: a Randomized Control Study
Brief Title: Real-time Sonography in Detecting Inadvertent Esophageal Intubation Among Difficult Intubation Patients
Acronym: SDEIDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Tian Yuan, MD, Physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PUMCH-ULT&ETT-DI
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication; Ultrasonography; Diagnostic Imaging
Keywords: Ultrasonography; Intubation; Intratracheal; Esophageal intubation; Difficult intubation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonography + direct visualization (Active Comparator): To detect using ultrasonography assisted direct visualization.
  Interventions: Procedure: Ultrasonography; Procedure: Direct visualization
- Direct visualization (Experimental): To detect using direct visualization.
  Interventions: Procedure: Direct visualization

INTERVENTIONS:
Procedure: Ultrasonography — The transducer will be placed over the anterior neck just above the suprasternal notch, in the transverse orientation. The position of the transducer could be adjusted to visualize both the esophagus and trachea. It will be considered as esophageal intubation if esophageal dilation or "double-tract" sign are noted.
  Arms: Ultrasonography + direct visualization
Procedure: Direct visualization — While performing the intubation, the intubator will report ETI if visualizing the tracheal tube passing through the glottis. Otherwise, it will be regarded as esophageal intubation.

SUMMARY:
Early detection of esophageal intubation, one of the most common complications while performing endotracheal intubation (ETI), is crucial to adequate airway management, especially among patients suspected of difficult intubation (DI). Detective approaches with ventilation require time, increase the risk of emesis and aspiration to patients, and increase the risk of particle aerosolization to health providers under the epidemic of aerosol-borne diseases. Our study will determine the effectiveness of real-time sonography assisted to direct visualization to detect esophageal intubation before ventilation among DI patients.

DETAILED DESCRIPTION:
A single-blind, superiority, randomized controlled study. 224 eligible participants requiring elective orotracheal intubation under general anesthesia with suspected DI will be randomized 1:1 to sonography and direct visualization versus direct visualization alone. The primary objective will be to investigate, in suspected DI patients, if the real-time sonography-assisted with direct visualization results in improved specificity in the detection of inadvertent esophageal intubation before ventilation compared with direct visualization while performing intubation. The secondary objectives will be to compare the sensitivity, positive likelihood ratio (LR+), negative likelihood ratio (LR-), diagnostic odds ratio (DOR), positive predictive value (PPV), negative predictive value (NPV), and detective self-confidence grade using sonography-assisted direct visualization vs direct visualization. Test characteristics will be calculated using standard formulas for a binomial proportion, and the corresponding 95% confidence intervals (CIs), by the Wilson interval method.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years old.
* Requiring elective orotracheal intubation under general anesthesia in the OR.
* Suspected DI according to airway assessments ，and with low risk of difficult ventilation.
* Planning to use a Macintosh laryngoscope blade on the first attempt, whether direct or video laryngoscopy.
* Signed written informed consent.
* Willingness for the primary anesthesia team to participate.

Exclusion Criteria:

* Anterior neck lesions, masses, lacerations, or subcutaneous emphysema.
* A history of neck operation or tracheotomy.
* Allergies to ultrasound coupling gel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
The specificity. | Upon or within three minutes of performing intubation.
  The detected negative/ true negative. According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In group ultrasonography assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.

SECONDARY OUTCOMES:
The sensitivity. | Upon or within three minutes of performing intubation.
  The detected positive/ true positive. According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In the group using ultrasonography-assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.
The positive likelihood ratio. | Upon or within three minutes of performing intubation.
  The positive likelihood ratio is calculated as sensitivity/(1 - specificity). According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In the group using ultrasonography-assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.
The negative likelihood ratio. | Upon or within three minutes of performing intubation.
  The negative likelihood ratio is calculated as (1 - sensitivity)/specificity. According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In the group using ultrasonography-assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.
The diagnostic odds ratio. | Upon or within three minutes of performing intubation.
  Positive likelihood ratios/Negative likelihood ratio. According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In the group using ultrasonography-assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.
The positive predictive value. | Upon or within three minutes of performing intubation.
  Cases of true positive among detective positive/ cases of detective positive. According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In the group using ultrasonography-assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.
The negative predictive value | Upon or within three minutes of performing intubation.
  Cases of true negative among detective negative/ cases of detective negative. According to the purpose of the proposed study, we will define esophageal intubation as positive, and endotracheal intubation as negative. In group direct visualization, positive and negative are defined as absent and present visualization of the tracheal tube passing through the glottis, respectively. In the group using ultrasonography-assisted direct visualization, positive is defined as sonography detection of esophageal dilation or "double-tract" sign, and negative is defined as direct visualization of the tracheal tube passing through the glottis. If neither the specific US nor the clear visualization is noted, the intubator and the sonographer will discuss and reach a consistent conclusion in three seconds.
The detective self-confidence grade | Upon or within three minutes of performing intubation.
  The detective self-confidence grade will be provided on a four-point scale of 1=" unsure", 2=" less sure", 3=" quite sure", and 4=" sure".

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Tian, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gottlieb M, Holladay D, Burns KM, Nakitende D, Bailitz J. Ultrasound for airway management: An evidence-based review for the emergency clinician. Am J Emerg Med. 2020 May;38(5):1007-1013. doi: 10.1016/j.ajem.2019.12.019. Epub 2019 Dec 11. PMID 31843325
- [Background] Brown CA 3rd, Bair AE, Pallin DJ, Walls RM; NEAR III Investigators. Techniques, success, and adverse events of emergency department adult intubations. Ann Emerg Med. 2015 Apr;65(4):363-370.e1. doi: 10.1016/j.annemergmed.2014.10.036. Epub 2014 Dec 20. PMID 25533140
- [Background] Das SK, Choupoo NS, Haldar R, Lahkar A. Transtracheal ultrasound for verification of endotracheal tube placement: a systematic review and meta-analysis. Can J Anaesth. 2015 Apr;62(4):413-23. doi: 10.1007/s12630-014-0301-z. Epub 2014 Dec 24. PMID 25537734